CLINICAL TRIAL: NCT04888572
Title: Assessment of the Association Between the New "Implant Disease Risk Assessment" Tool and Peri-implantitis or Implant Loss: a 5-year Retrospective Cohort Study.
Brief Title: Evaluation of the Novel Implant Disease Risk Assessment : a Retrospective Study (IDRA)
Acronym: IDRA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Tamara Rbeiz, Doctor of Dental Surgery, Saint-Joseph University
Other Study IDs: FMDA5/21
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Peri-Implantitis; Implant Expulsion
Keywords: Risk assessment; Risk factors; IDRA; Risk indicators; Peri-implantitis; Implant loss; Periodontal susceptibility
MeSH Terms: conditions — Peri-Implantitis | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Peri-Apical X-ray — Using a PCP UNC 15 Hu Friedy® periodontal probe and a gentle horizontal sweeping motion through the peri-implant "tunnel" or sulcus the examiner will assess bleeding on probing, the main factor in determining peri-implant inflammation and subsequently possible peri-implantitis. Then, using the same instrument, the author will examine whether there is an increase in the values of pocket depths compared to the initial values, highlighting an installation of peri-implant disease. Radiographically, evidence of bone loss after healing through taking a digital x-ray that will be viewed on DBSWIN® software will help authors make a diagnosis of peri-implantitis as well. It will be required that the digital film be perfectly parallel to the axis of the implant and the X-ray tube perpendicular to them in order to have an orthogonal radiograph.
  Other Names: Periodontal Probing

SUMMARY:
Given the novelty of this risk assessment tool, this study will be interested in evaluating its effectiveness through a retrospective approach. The IDRA risk will be analyzed at the time of loading the implant (s) in patients who have already placed an implant (s) during the last five years at the Department of Periodontology and Oral Surgery using the information collected from the periodontal file previously completed. Therefore, patients whose IDRA has been calculated will be called for a clinical and radiological examination to verify the development or not of peri-implantitis or the loss of the implant. In this way, this tool for predicting peri-implant disease will be evaluated to see if it is really effective.

DETAILED DESCRIPTION:
First, the files of patients who have placed an implant(s) at the Departments of Periodontology and Oral Surgery of the Faculty of Dental Medicine of Saint Joseph University, Beirut-Lebanon over the past five years (2015, 2016, 2017, 2018 and 2019) will be collected. Subsequently, thanks to the periodontal file and to the X-rays previously taken, the eight periodontal parameters necessary for the determination of the IDRA will be recorded (history of periodontitis; percentage of bleeding on probing; the number of teeth / implants with a pocket depth ≥ 5mm; the ratio between the level of bone loss (evaluated radiographically using retro-alveolar or panoramic X-rays already present in the patient's radiological record on the DBSWIN® software) and the patient's age ( at the time of loading the implant); the susceptibility to periodontitis (diagnosis) as described by the new classification of periodontal diseases and peri-implant from the World Workshop in 2017; compliance with maintenance visits; the distance (in mm) between the limit of the prosthesis and the marginal bone level (seen on the X-ray of the infrastructure or after sealing / screwing the prosthesis); prosthetic factors (such as the precision of adaptation of the prosthesis to the implant or the excess cement) and filled in on an Excel sheet. These data will then be reported online by following this link http://www.ircohe.net/IDRA which will make it possible to calculate by itself the IDRA of each patient.

As a result, each patient will have a personalized IDRA chart and they will be either at low, medium or high risk of developing peri-implantitis.

The retrospective analysis of the files being completed, the patients will be called to come to the Department of Periodontology in order to take the necessary measures to verify the presence or absence of a possible peri-implantitis on the one hand or the loss of the implant on the other hand.

ELIGIBILITY:
Inclusion Criteria:

1. Adults> 18 years old.
2. Patients who have placed one or more implants in the last five years at the Departments of Periodontology or Oral Surgery of the FMD and the implants have / have been loaded.
3. Patients whose periodontal file has been completed and the periodontal parameters required for IDRA reported.
4. Patients having an x-ray with the loaded implant or an x-ray during the try-in of the infrastructure.

Exclusion Criteria:

1. Patients with incomplete periodontal charts and missing parameters related to IDRA.
2. Patients not having an x-ray after loading the implant or during the try-in of the infrastructure
3. Totally edentulous patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients having placed one or more implants in the Departments of Periodontology or Oral Surgery between 01/01/2015 and 12/31/2019 and whose inclusion criteria are present to allow them to join the study .
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Association between IDRA and peri-implantitis | Up to thirty minutes
  To assess the association between the new risk measurement tool (IDRA) in patients with one or more implants and peri-implantitis Translation results To assess the association between the new risk measurement tool (IDRA) in patients with one or more implants and peri-implantitis.

SECONDARY OUTCOMES:
Association between IDRA and implant loss | Up to thirty minutes
  To assess the association between the new risk measurement tool (IDRA) in patients with one or more implants and loss of the implant.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Rebeiz, DentalSurg, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
The IPD that will be collected are confined to the Saint Joseph University's patients and their file are confidential.

REFERENCES:
- [Background] Heitz-Mayfield LJA, Heitz F, Lang NP. Implant Disease Risk Assessment IDRA-a tool for preventing peri-implant disease. Clin Oral Implants Res. 2020 Apr;31(4):397-403. doi: 10.1111/clr.13585. Epub 2020 Feb 20. PMID 32003037
- [Derived] Rebeiz T, Nasr L, Kassir AR, Menassa G, Chakar C. Assessment of the association between the Implant Disease Risk Assessment (IDRA) tool and peri-implantitis: a retrospective cohort study with up to 8 years of follow-up. Int J Oral Maxillofac Surg. 2024 Oct;53(10):845-852. doi: 10.1016/j.ijom.2024.05.002. Epub 2024 May 27. PMID 38806315
- See also: This website will allow the calculation of the IDRA of each patient — http://www.ircohe.net/IDRA